CLINICAL TRIAL: NCT01415375
Title: Prostate Cancer Education in African American Men
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: R01CA104223 (NIH)
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Prostate Cancer Screening Decision
Keywords: prostate-specific antigen (146-154); prostate-specific antigen (154-163)
MeSH Terms: interventions — Fruit

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prostate Cancer Screening Education (Experimental): Men in the experimental intervention group received an educational pamphlet on prostate cancer testing as well as tailored telephone education in which the interventionist provided information, answered questions, and conducted a values clarification exercise with the participant.
  Interventions: Behavioral: Prostate Cancer Screening Education
- Fruit and Vegetable Intake Education (Other): Men in the attention control group received an educational pamphlet on daily recommended servings of fruits and vegetables as well as tailored telephone education in which the interventionist provided information, answered participant's questions, and discussed any barriers to eating fruits and vegetables.
  Interventions: Behavioral: Fruit and Vegetable Intake Education

INTERVENTIONS:
Behavioral: Prostate Cancer Screening Education — tailored telephone education on prostate cancer testing
  Arms: Prostate Cancer Screening Education
Behavioral: Fruit and Vegetable Intake Education — tailored telephone education about fruit and vegetable consumption
  Arms: Fruit and Vegetable Intake Education

SUMMARY:
This study evaluates the efficacy of a tailored telephone intervention to promote informed decision making about prostate cancer testing among predominantly immigrant black men.

DETAILED DESCRIPTION:
African American and African-Caribbean men have the greatest prostate cancer incidence and mortality rate. Professional organizations provide conflicting recommendations regarding prostate cancer testing but generally agree that men learn about the risks and benefits of testing and share in decisions about testing based on their personal preferences. This study was designed to assess the effects of a decision support intervention on men's knowledge about prostate cancer testing, participation in medical decisions about testing, decision conflict related to testing, and the congruence between prostate cancer testing intentions and behaviors. A randomized controlled trial was conducted. Participants were randomized into one of two conditions: (a) tailored telephone education about prostate cancer testing (intervention group) or (b) tailored telephone education about national guidelines for fruit and vegetable consumption (attention control group).

ELIGIBILITY:
Inclusion Criteria:

* 45 to 70 year old
* African descent
* accessible by telephone
* have primary care physician

Exclusion Criteria:

* Prostate cancer test in 12 months prior to enrollment
* History of prostate cancer

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2004-09; Primary Completion 2007-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
congruence between prostate cancer testing intention and behavior | 1 and 2 years post randomization
  Congruence between men's stated intentions to get tested and their actual testing behavior, validated by medical claims at 1 and 2 year follow-up. Intention-behavior agreement was coded as congruent (1), whereas disagreement was coded as incongruent (0).
Knowledge about prostate cancer and prostate cancer tests | baseline and 8 months post randomization
  12 item knowledge index with questions on testing, risk factors and epidemiology, and treatment effectiveness and side effects. Percent correct was used as the outcome measure.
Decisional conflict | 8 months post randomization
  Used a modified version of the 16 item Decisional Conflict Scale with the 3 level response category suggested for low literacy populations.
Verified doctor visit to discuss prostate cancer testing | 2 years post randomization
  Visit with physician to talk about prostate cancer testing, with visit verified through medical claims records

SECONDARY OUTCOMES:
State anxiety | baseline and 8 months post-randomization
  Used a 7 item subscale of the Hospital Anxiety and Depression Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lepore, PhD, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Lepore SJ, Wolf RL, Basch CE, Godfrey M, McGinty E, Shmukler C, Ullman R, Thomas N, Weinrich S. Informed decision making about prostate cancer testing in predominantly immigrant black men: a randomized controlled trial. Ann Behav Med. 2012 Dec;44(3):320-30. doi: 10.1007/s12160-012-9392-3. PMID 22825933